CLINICAL TRIAL: NCT02936700
Title: Identification of Prognostic Biomarkers by fMRI of Acceptance and Commitment Therapy in Suicidal Behavior Disorder
Brief Title: Biomarkers of Efficiency of Acceptance and Commitment Therapy in Suicidal Behavior
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UF 9519; 2014-A01781-46 (Other: Agence Nationale de Sécurité des Médicaments)
Record Dates: First submitted 2016-07-15; First posted 2016-10-18 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Actual Suicidal Behavior Disorder
Keywords: Psychiatry; Suicide; Randomized controlled trial; ACT; fMRI
MeSH Terms: conditions — Suicide | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Other): Add on relaxation group
  Interventions: Behavioral: Relaxation
- Therapy ACT (Experimental): Add on ACT group
  Interventions: Behavioral: ACT therapy

INTERVENTIONS:
Behavioral: Relaxation — relaxation program consists of 7 weekly, 2 hours sessions led by two therapist. Each group will consist of 7 participants.
  Arms: Control group
Behavioral: ACT therapy — 7 weekly, 2 hours sessions led by two therapist. Each group will consist of 7 participants. The ACT program aims at
  * decreasing the tendency to try to escape unpleasant mental experiences
  * increasing psychological flexibility
  * developing acceptance of psychological events and engagement in valued actions
  Arms: Therapy ACT

SUMMARY:
Suicidal behaviors (SB) are a major health problem in France:10,000 suicides and 220,000 suicide attempts every year. SB management is therefore a major public health issue. Recently, investigators have demonstrated the interest of acceptance and commitment therapy (ACT) as an add-on treatment to reduce intensity and severity of suicidal ideation in depressed patients having a history of suicide attempt within previous year (i.e actual SB disorder according to the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5)). Based on structural and functional findings, it is admitted orbitofrontal and ventral prefrontal cortices play a role in suicidal vulnerability. Interestingly, previous functional MRI (fMRI) studies have also reported the modulation of these regions by ACT in subjects suffering from chronic pain. fMRI could thus be an interesting tool to identify biomarkers of SB and its improvement by ACT.

The aim of study is to investigate neural biomarkers of ACT efficiency in patients with SB disorder. Patients having a history of SB within previous year were randomized in an ACT program (21 patients) or relaxation program (21 patients) during 7 weeks. Before and after the completion of the group, they performed 3 tasks during fMRI: implicit emotional visualization, Cyberball game, motivational task Investigators will compare cerebral activations between groups, between pre and post intervention as well as measure baseline cerebral activations associated with improvement of suicidal ideation during follow up.

DETAILED DESCRIPTION:
42 patients having a history of suicide attempt within the year preceding inclusion have been recruited.

First visit or inclusion (within 2 weeks preceding the beginning of the program): clinical, biological assessment and fMRI acquisition Second visit (within 2 weeks +/- 1 week following completion of the program): clinical assessment and fMRI acquisition Third visit (within 3 months +/- 2 weeks following completion of the program): clinical assessment

ELIGIBILITY:
Inclusion criteria:

* Between 18 and 65 years
* Having signed informed consent
* Main diagnosis of major depressive episode (DSM-5 criteria)
* History of suicide attempt within the year
* Able to understand nature, aims, methodology of the study and agree to cooperate in clinical, radiological assessments.

Exclusion criteria:

* Current diagnosis of substance abuse or dependence in the last 6 months (including tobacco and alcohol)
* Current lifetime diagnosis of schizophrenia, or schizoaffective disorder
* Current diagnosis of manic, hypomanic according to DSM-5 criteria
* Contraindications for the use of MRI, : metallic artificial heart valve, pacemaker, ferromagnetic cerebrovascular clips, metallic foreign body including brain mobilized or intraocular ferromagnetic prosthesis impossibility of absolute immobility, claustrophobia.
* Lifetime history of traumatic brain injury with loss of consciousness
* Pregnancy
* Patient on protective measures (guardianship or trusteeship)
* Patient for which the maximum annual amount of allowances 4 500 euros has been reached

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-09-05 (Actual); Study Completion 2017-03-05 (Actual)

PRIMARY OUTCOMES:
Variation of cerebral activation when viewing angry versus neural faces during an implicit emotional visualization task | At 2 weeks after group completion
  Comparison between inclusion and 2 weeks after group completion of cerebral activation within ACT group
Variation of cerebral activation when viewing angry versus neural faces during an implicit emotional visualization task | At 2 weeks after group completion
  Comparison between inclusion and 2 weeks after group completion of cerebral activation within relaxation group
Baseline activation when viewing angry vs. neutral faces during an implicit emotional visualization task | At 3 months after therapy
  comparison between subjects with suicidal ideation vs. without suicidal ideation at 3 months after therapy

SECONDARY OUTCOMES:
Activation of specific brain regions when viewing sad, happy and disgust faces versus neutral faces during an implicit emotional visualization task | At the inclusion, and 2 weeks after the end of the therapy
  comparison between the two groups and before/after therapy / Association between baseline activation and improvement of suicidal ideation
Activation of specific brain regions during Cyberball game, a validated exclusion task | At the inclusion, and 2 weeks after the end of the therapy
  comparison between the two groups and before/after therapy / Association between baseline activation and improvement of suicidal ideation
Activation of specific brain regions during a motivational task | At the inclusion, and 2 weeks after the end of the therapy
  comparison between the two groups and before/after therapy / Association between baseline activation and improvement of suicidal ideation
Change of activation of default mode network (DMN) during resting state acquisition | Baseline acquisition and 2 weeks after therapy
  Comparison between groups
Baseline activation of DMN during resting state acquisition | Baseline acquisition and clinical assessment at 3 months after therapy
  Comparison between subjects with suicidal ideation versus without at 3 months after therapy
Baseline fraction of anisotropy | Baseline acquisition and clinical assessment at 3 months
  Comparison between subjects with suicidal ideation versus without at 3 months after therapy
Evolution of suicidal ideation measured by the Columbia Suicide Severity Rating Scale (CSSRS) | At the inclusion, 2 weeks after the end of the therapy and 3 months after the end of the therapy
  Comparison between the beginning and the end within each group and comparison between the two groups
Evolution of depressive state during the follow up measured by the Inventory of Depressive Symptomatology (IDSC-30) | At the inclusion, 2 weeks after the end of the therapy and 3 months after the end of the therapy
  Comparison between the beginning and the end within each group and comparison between the two groups
Evolution of psychologic pain during the follow up | At the inclusion, 2 weeks after the end of the therapy and 3 months after the end of the therapy
  Comparison between the beginning and the end within each group and comparison between the two groups by Likert scale
Evolution of anger during the follow up. | At the inclusion, 2 weeks after the end of the therapy and 3 months after the end of the therapy
  Comparison between the beginning and the end within each group and comparison between the two groups by the STAXI scale (Spielberger State-Trait Anger Expression Inventory)
Evolution of clinical global impression during the follow up. | At the inclusion, 2 weeks after the end of the therapy and 3 months after the end of the therapy
  Comparison between the beginning and the end within each group and comparison between the two groups by the CGI (Clinical Global Impressions scale)
Evolution of suicidal ideation measured by the Scale for Suicide Ideation (SSI) | At the inclusion, 2 weeks after the end of the therapy and 3 months after the end of the therapy
  Comparison between the beginning and the end within each group and comparison between the two groups
Evolution of depressive state during the follow up measured by the Quick Inventory of Depressive Symptomatology (QIDS-RS) | At the inclusion, 2 weeks after the end of the therapy and 3 months after the end of the therapy
  Comparison between the beginning and the end within each group and comparison between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier Hospital University, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617